CLINICAL TRIAL: NCT00002031
Title: Evaluation of the Epidermal Langerhans Cell Population in AIDS / ARC Patients by the Topical Application of a Potent Contact Allergen (1-Chloro-2,4-Dinitro-Chlorobenzene) (DNCB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 047A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: HIV Infections
Keywords: Langerhans Cells; Dinitrochlorobenzene; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Dinitrochlorobenzene

INTERVENTIONS:
Drug: Dinitrochlorobenzene

SUMMARY:
To evaluate the effect of application of Dinitrochlorobenzene (DNCB) on the number, morphology, and antigen expression of epidermal Langerhans cells in AIDS and AIDS related complex (ARC) patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Stage III or IV HIV infection.
* Provide informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Kaposi's sarcoma lesions in the proposed treatment sites.
* Liable to require radiation or chemotherapy during the course of the study.
* Not likely to survive the length of the study.
* Obvious ultra-violet-irradiated skin damage in the treatment areas and anyone with recent UV exposure or likely to have such exposure (e.g.:
* holiday tans obtained in Hawaii, members of UV box tanning salons, etc.) Allergy to lidocaine.

Concurrent Medication:

Excluded:

* Other Immunomodulators.

Concurrent Treatment:

Excluded:

* Radiation.

Patients with the following are excluded:

* Kaposi's sarcoma lesions in the proposed treatment sites.
* Liable to require radiation or chemotherapy during the course of the study.
* Not likely to survive the length of the study.
* Obvious ultra-violet-irradiated skin damage in the treatment areas.
* Allergy to lidocaine.

Prior Medication:

Excluded:

* Prior DNCB therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California, United States

REFERENCES:
- [Background] Stricker RB, Elswood BF. Dendritic cells and dinitrochlorobenzene (DNCB): a new treatment approach to AIDS. Immunol Lett. 1991 Aug;29(3):191-6. doi: 10.1016/0165-2478(91)90169-b. PMID 1769706